CLINICAL TRIAL: NCT01423604
Title: A Randomized Phase 2 Study of Ruxolitinib Efficacy and Safety in Combination With Capecitabine for Subjects With Recurrent or Treatment Refractory Metastatic Pancreatic Cancer (The RECAP Trial)
Brief Title: Study of Ruxolitinib in Pancreatic Cancer Patients
Acronym: RECAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18424-262
Record Dates: First submitted 2011-08-22; First posted 2011-08-26 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine and ruxolitinib (Experimental)
  Interventions: Drug: Capecitabine; Drug: Ruxolitinib
- Capecitabine and placebo (Placebo Comparator)
  Interventions: Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: Capecitabine — Capecitabine starting dose - 2000 mg/m^2 (1000 mg/m^2 twice a day (BID)) (NOTE: Frequency of administration may be adjusted during the study.)
Drug: Ruxolitinib — Ruxolitinib starting dose - 15 mg BID (NOTE: Starting dose of randomized study drug may be 10 mg BID based on results from safety run-in study. Dose of ruxolitinib may be increased during randomized study.)
  Arms: Capecitabine and ruxolitinib
Drug: Placebo — Placebo matching ruxolitinib
  Arms: Capecitabine and placebo

SUMMARY:
The purpose of this study was to determine whether ruxolitinib added to capecitabine is effective in improving the overall survival of patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The study consisted of an open-label, safety run-in period that was composed of 1 patient cohort with 9 patients/cohort. This phase of the study determined the safety of the capecitabine/ruxolitinib combination in this patient population.

A randomized, double-blind study with two treatment arms was conducted once the safety run-in results from the first part of the study showed that the capecitabine/ruxolitinib combination was safe and additional patients could be treated. All patients have received capecitabine therapy in addition to the ruxolitinib or placebo (Study Drug).

Treatment for all patients consisted of repeating 21-day cycles. Capecitabine was self-administered for the first 14 days of each cycle, and the Study Drug was self-administered during the entire 21-day cycle. Treatment cycles continued as long as the regimen was tolerated and the patient did not meet any of the discontinuation criteria. In the event of disease progression, capecitabine therapy was discontinued but the Study Drug could continue to be administered. Subjects who discontinued treatment with the Study Drug continued to be followed to obtain information regarding subsequent treatment regimens and survival.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of metastatic pancreatic cancer; subjects must have had measurable, or evaluable disease that was histologically confirmed
* Karnofsky performance status of ≥ 60
* Subjects must have failed 1st-line gemcitabine treatment for metastatic pancreatic cancer:

  o An alternate chemotherapeutic agent was an acceptable substitute as 1st-line therapy in the event that the subject was intolerant to or ineligible to receive gemcitabine
* ≥ 2 weeks elapsed from the completion of previous chemotherapy, and subjects must have recovered or been at new stable baseline from any related toxicities

Exclusion Criteria:

* More than 1 prior chemotherapy regimen (not including adjuvant therapy) for metastatic disease
* Evidence of central nervous system (CNS) metastases (unless stable for > 3 months) or history of uncontrolled seizures
* Ongoing radiation therapy or prior radiation therapy administered as a second-line treatment
* Other active malignancy except basal or squamous carcinoma of the skin
* Inability to swallow food or any condition of the upper GI tract that precluded administration of oral medications
* Inadequate renal, hepatic and bone marrow function demonstrated by clinical observations and/or laboratory assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Williams, MD, Study Director — Incyte Corporation
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Burbank, California
  - Los Angeles, California
  - Santa Monica, California
  - Denver, Colorado
  - Stamford, Connecticut
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Arlington Heights, Illinois
  - Elks Grove Village, Illinois
  - Indianapolis, Indiana
  - Sioux City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Novi, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Lake Success, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Canton, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Danville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Knoxville, Tennessee
  - San Antonio, Texas
  - Richmond, Virginia
  - Green Bay, Wisconsin

REFERENCES:
- [Derived] Hurwitz HI, Uppal N, Wagner SA, Bendell JC, Beck JT, Wade SM 3rd, Nemunaitis JJ, Stella PJ, Pipas JM, Wainberg ZA, Manges R, Garrett WM, Hunter DS, Clark J, Leopold L, Sandor V, Levy RS. Randomized, Double-Blind, Phase II Study of Ruxolitinib or Placebo in Combination With Capecitabine in Patients With Metastatic Pancreatic Cancer for Whom Therapy With Gemcitabine Has Failed. J Clin Oncol. 2015 Dec 1;33(34):4039-47. doi: 10.1200/JCO.2015.61.4578. Epub 2015 Sep 8. PMID 26351344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The open-label, safety run-in (1 cohort) was designed to confirm the safety of the combination of ruxolitinib and capecitabine in subjects with advanced or metastatic adenocarcinoma of the pancreas. The double-blind portion was 2 treatment groups randomized 1:1: ruxolitinib plus capecitabine or matching placebo plus capecitabine.
Groups:
- Ruxolitinib: Part 1: Subjects received capecitabine 2000 mg/m^2 (1000 mg/m^2 twice a day (BID)) + ruxolitinib 15 mg BID.
  Part 2: Subjects received ruxolitinib 15 mg BID plus capecitabine at a starting dose of 2000 mg/m^2 (1000 mg/m^2 twice a day [BID]).
- Placebo: Part 2: Matching placebo tablets were administered as oral doses in the same manner as active drug during the randomized portion of the study. Capecitabine starting dose - 2000 mg/m^2 (1000 mg/m^2 twice a day [BID]).
Period: Safety Run-In
Arm/Group | Ruxolitinib | Placebo
Started | 9 | 0
Completed | 0 | 0
Not Completed | 9 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Disease progression | 3 | 0
Not completed — Patient decision | 1 | 0
Period: Randomized
Arm/Group | Ruxolitinib | Placebo
Started | 64 | 63
Completed | 1 (As of 07August2015, 1 subject was receiving treatment in the randomized portion.) | 0
Not Completed | 63 | 63
Not completed — Adverse Event | 4 | 10
Not completed — Death | 1 | 0
Not completed — Physician Decision | 16 | 13
Not completed — Other - unspecified | 37 | 31
Not completed — Patient decision | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Ruxolitinib - Safety Run-In: Subjects received capecitabine 2000 mg/m^2 (1000 mg/m^2 twice a day [BID]) + ruxolitinib at 15 mg BID.
- Ruxolitinib: Subjects received ruxolitinib 15 mg BID plus capecitabine at a starting dose of 2000 mg/m^2 (1000 mg/m^2 twice a day [BID]).
- Placebo: Matching placebo tablets were administered as oral doses in the same manner as active drug during the randomized portion of the study. Capecitabine starting dose - 2000 mg/m^2 (1000 mg/m^2 twice a day [BID]).
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib - Safety Run-In | Ruxolitinib | Placebo | Total
Number analyzed (Participants) | 9 | 64 | 63 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.4) | 65.7 (9.3) | 66.3 (9.8) | 66.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 23 | 29 | 57
  Male | 4 | 41 | 34 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 5 | 6
  Not Hispanic or Latino | 9 | 62 | 58 | 129
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 9 | 6 | 18
  White | 5 | 54 | 54 | 113
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Height [Mean (Standard Deviation); unit: cm] — Treatment Group Ruxolitinib (N = 60); Placebo (N = 60)
  cm | 171.67 (14.11) | 171.29 (11.93) | 168.27 (10.25) | 169.78 (11.18)
Weight [Mean (Standard Deviation); unit: kg] — Treatment Group Ruxolitinib (N = 60); Placebo (N = 60)
  kg | 75.051 (17.317) | 75.014 (21.914) | 69.299 (16.260) | 72.156 (19.427)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Treatment Group Ruxolitinib (N = 60); Placebo (N = 60)
  kg/m^2 | 25.3 (4.209) | 25.354 (6.332) | 24.243 (4.237) | 24.789 (5.394)
Body surface area [Mean (Standard Deviation); unit: m^2] — Treatment Group Ruxolitinib (N = 60); Placebo (N = 60)
  m^2 | 1.869 (0.287) | 1.863 (0.297) | 1.791 (0.248) | 1.827 (0.275)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was measured as the length of time (in days) between the randomization date and the date of death.
Time Frame: Primary analysis includes study data from the start of the study (first dose for that subject) until the death of the subject (up to 8 months).
Population: The intent-to-treat (ITT) population included subjects randomized in Part 2 of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 64 | 63
days | 136.5 [95.0 to 196.0] | 129.5 [71.0 to 179.0]
Statistical Analysis 1: Comparison: Ruxolitinib vs Placebo; Test type: Superiority or Other; p = 0.0494, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.733, 95% CI 2-sided [0.506 to 1.061]
Statistical Analysis 2: Comparison: Ruxolitinib vs Placebo; Cox Regression Analysis of Overall Survival: C-reactive protein (CRP) > 13 μg/ml; Statistical analysis plan (SAP) specified subgroup analysis; Test type: Superiority or Other; p = 0.0081, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.502, 95% CI 2-sided [0.281 to 0.888]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the length of time between the date of randomization and the earlier of death or progressive disease (PD), whichever was earlier, as assessed by RECIST. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Analysis includes study data from the start of the study (first dose for that subject) until death or PD, whichever was earlier up to 8 months.
Population: The intent-to-treat (ITT) population included subjects randomized in Part 2 of the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 64 | 63
days | 51.0 [42.0 to 84.0] | 46.0 [41.0 to 70.0]
Statistical Analysis 1: Comparison: Ruxolitinib vs Placebo; Test type: Superiority or Other; p = 0.1340, Cox proportional hazards model — Two-sided p-value; Efron approximation of hazard ratio = 0.750, 95% CI 2-sided [0.513 to 1.094]

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) was defined as the percentage of participants with either a confirmed complete response (CR) or partial response (PR) measured by the investigator per modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 criteria during the treatment period. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Measured every 4 weeks for duration of study treatment (up to 8 months)
Population: The intent-to-treat (ITT) population included subjects randomized in Part 2 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 64 | 63
percentage of participants
  Overall response | 7.8 | 1.6
  Complete response | 1.6 | 0.0
  Partial response | 6.3 | 1.6

4. Secondary Outcome: Durable Response Rate
Description: Durable response was defined as subjects with a response of Partial response (PR) or better at 2 subsequent measurements that were at least 4 weeks apart.
Time Frame: Measured every 4 weeks until death or PD, whichever was earlier (up to 8 months)
Population: The intent-to-treat (ITT) population included subjects randomized in Part 2 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 64 | 63
percentage of participants | 7.8 | 0.0
Statistical Analysis 1: Comparison: Ruxolitinib vs Placebo; Test type: Superiority or Other; p = 0.0236, Pearson's chi-square test

5. Secondary Outcome: Summary of Clinical Benefit
Description: A subject was considered a clinical benefit responder if he/she met at least 1 of the following criteria:
  1. Subject showed improvement in at least one of the following parameters on successive scheduled observations without worsening in the others: pain intensity, analgesic use, or performance status
  2. Subject was stable or improved on the pain intensity, analgesic use, and performance status and had a ≥ 7% increase in body weight maintained for 2 consecutive reporting periods that was not because of fluid accumulation.
Time Frame: Measured every 4 weeks until death or PD, whichever was earlier (up to 8 months)
Population: The intent-to-treat (ITT) population included subjects randomized in Part 2 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 64 | 63
percentage of participants
  Subjects with clinical benefit | 12.5 | 1.6
  Pain intensity - Improved | 10.9 | 1.6
  Analgesic use - Improved | 4.7 | 0.0
  Karnofsky performance status - Improved | 3.1 | 0.0
  Body weight - Improved | 3.1 | 0.0

ADVERSE EVENTS:
Time Frame: From the start of the study (first dose for that subject) until the end of the Adverse Event (AE) period (30 days after the last dose) or death, whichever was earlier (up to 8 months).
Description: Safety evaluable population included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Ruxolitinib (Safety Run-In): Subjects received capecitabine 2000 mg/m^2 daily (taken as 1000 mg/m2 twice daily [BID]) + ruxolitinib 15 mg BID
Arm/Group | Ruxolitinib (Safety Run-In) | Ruxolitinib | Placebo
Serious Adverse Events (participants affected / at risk) | 5/9 | 32/59 | 35/60
Other Adverse Events (participants affected / at risk) | 9/9 | 57/59 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (Safety Run-In) (N=9) | Ruxolitinib (N=59) | Placebo (N=60)
Anemia (Blood and lymphatic system disorders) | 0 | 4 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Cardiorespiratory arrest (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 5
Ascites (Gastrointestinal disorders) | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Fecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Necrotizing colitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 1
Asthenia (General disorders) | 1 | 0 | 2
Device occlusion (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 5 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Klebsiella bacteremia (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 4
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
International normalized ratio increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Colostomy (Surgical and medical procedures) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Prothrombin Time Prolonged (Investigations) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (Safety Run-In) (N=9) | Ruxolitinib (N=59) | Placebo (N=60)
Anemia (Blood and lymphatic system disorders) | 7 | 30 | 12
Fatigue (General disorders) | 2 | 29 | 26
Abdominal pain (Gastrointestinal disorders) | 5 | 22 | 23
Diarrhea (Gastrointestinal disorders) | 4 | 22 | 17
Nausea (Gastrointestinal disorders) | 4 | 21 | 27
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 19 | 19
Stomatitis (Gastrointestinal disorders) | 3 | 16 | 8
Vomiting (Gastrointestinal disorders) | 5 | 14 | 21
Decreased appetite (Metabolism and nutrition disorders) | 2 | 12 | 20
Dehydration (Metabolism and nutrition disorders) | 5 | 12 | 10
Constipation (Gastrointestinal disorders) | 2 | 11 | 19
Pyrexia (General disorders) | 1 | 10 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 12
Asthenia (General disorders) | 2 | 7 | 8
Dizziness (Nervous system disorders) | 1 | 7 | 5
Edema peripheral (Metabolism and nutrition disorders) | 3 | 7 | 6
Flatulence (Gastrointestinal disorders) | 1 | 7 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 6 | 7
Ascites (Gastrointestinal disorders) | 1 | 6 | 10
Hyponatremia (Metabolism and nutrition disorders) | 0 | 6 | 2
Hypotension (Vascular disorders) | 1 | 6 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 6 | 3
Pneumonia (Infections and infestations) | 0 | 6 | 3
Chills (General disorders) | 1 | 5 | 2
Confusional state (Psychiatric disorders) | 1 | 5 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 3
Weight decreased (Investigations) | 1 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Edema (Metabolism and nutrition disorders) | 2 | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 4 | 3
Candidiasis (Infections and infestations) | 1 | 3 | 4
Depression (Psychiatric disorders) | 0 | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 3 | 1
Hemorrhoids (Vascular disorders) | 0 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Insomnia (Psychiatric disorders) | 0 | 3 | 7
International normalized ratio increased (Investigations) | 1 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 3 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Somnolence (Psychiatric disorders) | 0 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 5
Headache (Nervous system disorders) | 0 | 2 | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Urinary tract infection (Renal and urinary disorders) | 2 | 2 | 7
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Bacteremia (Infections and infestations) | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 4
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Tongue pigmentation (Gastrointestinal disorders) | 1 | 0 | 0
Catheter site discharge (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Suprapubic pain (General disorders) | 1 | 0 | 0
Temperature Intolerance (General disorders) | 1 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Nail Bed Infection (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Open Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Prothrombin Time Prolonged (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Testicular Oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.